CLINICAL TRIAL: NCT04243720
Title: Immune Resistance Interrogation Study
Acronym: IRIS
Status: Recruiting | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: IRIS; CAPCR ID (Other: 19-6224)
Record Dates: First submitted 2020-01-20; First posted 2020-01-28 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Cancer; Solid Tumor; Metastatic Cancer; Immune Resistance
Keywords: Molecular Profiling; Liquid Biopsy; Tumor Biopsy; Circulation Tumor DNA; Epigenetics; Microbiome; Radiomics; Immune Analysis; Immunohistochemistry
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood samples collected serially for DNA extraction under the LIBERATE protocol.
  Archived tumor sample (if available) collected for DNA extraction. Fresh tumor biopsy sample (if available) collected for DNA extraction. Stool sample (if available) collected for DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Immune Resistance Interrogation Study (IRIS): Patients with a histological or cytological diagnosis of solid malignancies. Patients must have progressed on immunotherapy as their most recent line of therapy.

SUMMARY:
This is a prospective research study which will include patients who have progressed on immunotherapy as their most recent line of therapy. This study aims to characterize whether patients who fail to respond to immunotherapy versus patients who respond initially but after a period of time progress demonstrate different genomic, transcriptomic, epigenetic, immunophenotyping profiles. Patients will have a one-time fresh tumor biopsy. Serial blood samples (total amount of blood drawn may not exceed the lesser of 50 mL or 3 mL/kg in an 8 week period), archival tissue (if available) and one stool sample will be collected.

DETAILED DESCRIPTION:
Although there has been some success with the use of immunotherapy treatments specifically antibodies that block the programmed death 1 receptor (PD1/L1), the majority of cancer patients either fail to respond (primary resistance) or respond initially but progress after a period of time (acquired resistance) when treated with immunotherapy agents. The hypothesis being tested is whether patients who have primary versus acquired resistance to immunotherapy demonstrate different genomic, transcriptomic, immunophenotypic and/or epigenetic profiles.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a histological or cytological diagnosis of solid malignancies, with at least one tumor lesion amenable to core needle biopsy and consent to such a procedure.
* Patients must have progressed on immunotherapy (defined as anti-PD1/PD-L1 antibodies given as monotherapy or as part of a combination therapy) as their most recent line of therapy. Patients will be classified into two groups: 1) those who benefitted from immunotherapy with either complete response (CR), partial response (PR) or prolonged stable disease (SD) lasting at least 6 months with subsequent progression or who had disease progression after at least 12 weeks from the last dose of immunotherapy in the adjuvant setting (i.e. acquired resistance), 2) those whose disease is primary refractory to immunotherapy with disease progression at their first on-treatment imaging, those who benefitted from immunotherapy with stable disease (SD) but progressed in <6 months or those that had progressive disease earlier than 12 weeks from the last dose of immunotherapy in the adjuvant setting.
* Patients must be of good performance status, ECOG 0-1, for subsequent anticancer therapy, with either standard treatment or within the context of a clinical trial.
* Patients must be ≥ 18 years old.
* Patients must have provided voluntary written informed consent.

Exclusion Criteria:

* Any condition that could interfere with a patient's ability to provide informed consent such as dementia or severe cognitive impairment.
* Any contraindication to undergoing venipuncture.
* Any condition that, in the opinion of the Investigator, would interfere with patient safety, or evaluation of the collected specimens and interpretation of study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a diagnosis of solid tumor malignancy who progressed on immunotherapy as their most recent line of therapy.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-08-26 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Genomic changes associated with primary or acquired resistance to immunotherapy given alone or in combination in patients with advanced solid tumors | Through study completion, up to 4 years
  The genomic parameters for radiomic imaging analysis will be derived from patients' routine CT scans to study changes in radiomic signatures during treatment.
Transcriptomic changes associated with primary or acquired resistance to immunotherapy given alone or in combination in patients with advanced solid tumors | Through study completion, up to 4 years
  The transcriptomic parameters for radiomic imaging analysis will be derived from patients' routine CT scans to study changes in radiomic signatures during treatment.
Immunophenotypic changes associated with primary or acquired resistance to immunotherapy given alone or in combination in patients with advanced solid tumors | Through study completion, up to 4 years
  The immunophenotypic parameters for radiomic imaging analysis will be derived from patients' routine CT scans to study changes in radiomic signatures during treatment.
Epigenetic changes associated with primary or acquired resistance to immunotherapy given alone or in combination in patients with advanced solid tumors | Through study completion, up to 4 years
  The epigenetic parameters for radiomic imaging analysis will be derived from patients' routine CT scans to study changes in radiomic signatures during treatment.

SECONDARY OUTCOMES:
Genomic changes associated with subsequent anticancer therapies in patients with advanced solid tumors who have progressed on immunotherapy | Through study completion, up to 4 years
  The genomic parameters for radiomic imaging analysis will be derived from patients' routine CT scans to study changes in radiomic signatures during treatment.
Transcriptomic changes associated with subsequent anticancer therapies in patients with advanced solid tumors who have progressed on immunotherapy | Through study completion, up to 4 years
  The transcriptomic parameters for radiomic imaging analysis will be derived from patients' routine CT scans to study changes in radiomic signatures during treatment.
Immunophenotyping changes associated with subsequent anticancer therapies in patients with advanced solid tumors who have progressed on immunotherapy | Through study completion, up to 4 years
  The immunophenotypic parameters for radiomic imaging analysis will be derived from patients' routine CT scans to study changes in radiomic signatures during treatment.
Epigenetic changes associated with subsequent anticancer therapies in patients with advanced solid tumors who have progressed on immunotherapy | Through study completion, up to 4 years
  The epigenetic parameters for radiomic imaging analysis will be derived from patients' routine CT scans to study changes in radiomic signatures during treatment.

OTHER OUTCOMES:
Radiomic changes associated with primary or acquired resistance to immunotherapy given alone or in combination in patients with advanced solid tumors | Through study completion, up to 4 years
  Dynamic changes in radiomic signatures of tumors between commencement of systemic treatment and disease progression will be analysed from serial CT scans (normally performed at base line and approximately every 2-3 months thereafter until disease progression).
Radiomic changes associated with subsequent anticancer therapies in patients with advanced solid tumors who have progressed on immunotherapy | Through study completion, up to 4 years
  Tumor radiomic signatures will be used to study how phenotypic characteristics of tumors change during systemic therapy and how these signatures correlate with genomic, transcriptomic, immunophenotypic and epigenetic signatures
Fecal microbiome changes associated with primary or acquired resistance to immunotherapy given alone or in combination in patients with advanced solid tumors | Through study completion, up to 4 years
  DNA extraction will be performed and subjected to Shotgun sequencing. Bioinformatic analysis will be performed to determine microbial taxa composition (operation taxa units - OTU's) and diversity, including abundance plots at class, genus and species levels, alpha diversity (Rarefaction curve, Shannon curve, Rank Abundance curve) and beta diversity ((Un)weighted unifrac distance, PCoA) plots.

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, MD, Principal Investigator — Princess Margaret Cancer Centre; Anna Spreafico, MD, Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada